CLINICAL TRIAL: NCT03855592
Title: Observational Epidemiological Study of Cancer-associated Thrombosis: Registry of Thrombosis & NEoplasia of SEOM (TESEO Study)
Brief Title: Registry of Thrombosis & NEoplasia of "Sociedad Española de Oncología Médica"
Acronym: TESEO
Status: Recruiting | Type: Observational
Sponsor: Fundación Sociedad Española de Oncologia Médica (Other)
Responsible Party: Sponsor
Other Study IDs: SEOM-TESEO-2017-01
Record Dates: First submitted 2019-02-19; First posted 2019-02-27 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Thromboembolism; Cancer
MeSH Terms: conditions — Thromboembolism; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiological, observational, non-interventional, multicentric study on patients diagnosed with cancer who develop a venous or arterial thromboembolic episode, symptomatic or incidental, within a month prior to cancer diagnosis or at anytime after such diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age with a histologically confirmed diagnosis of malignant tumor.
* Venous or arterial thromboembolism episode, symptomatic or incidental, in the month prior or any time after the cancer diagnosis and in the three previous months to enrollment, confirmed with an imaging technique: Doppler echocardiography, computed tomography (CT) angiography, etc.
* Signing of informed consent.

Exclusion Criteria:

* Clinical diagnosis of thromboembolic event without radiological confirmation.
* Presenting a single episode of superficial thrombophlebitis without association with another thromboembolic event.
* Each patient will be recorded just once, and therefore a second thromboembolic event will be considered a rethrombosis and will be recorded as such. Patients with a rethrombosis and a previous thromboembolic event before the start of the study in each center will not be able to be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Location of origin of the thromboembolytic event | Baseline
  Distribution in the number of patients according to the anatomical location affected by the thromboembolytic event.
Vessel of origin of the thromboembolytic event | Baseline
  Distribution in the number of patients according to the type of vessel affected by the thromboembolytic event.
Thromboembolytic event diagnosis type | Baseline
  Proportion of patients with incidental versus symptomatic thormboembolic events
Primary tumor at the time of the thromboembolic event | Baseline
  Distribution of patients according to the organ affected by the primary tumor.
Tumor-Node-Metastasis classification | Baseline
  Based on the American Joint Committee on Cancer 2018 Tumor-Node-Metastasis classification system: T for extent or size of the tumor, N for lymph nodes spread and M for metastasis.
Time between cancer diagnosis and thromboembolic event | Baseline
  Based on date on confirmed diagnosis of cancer (primary tumor) and date of thromboembolic event
Patient situation at the last visit | 12 months
  Number of patients with rethrombosis, bleeding, other complications, tumor progression or death.
Characteristics of treatment administered for cancer | Baseline
  Based on the number of patients prescribed with chemotherapy, radiation therapy, hormonal therapy, erythropoietin, transfusions, surgery, catheter, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Muñoz, M.D., Study Chair — Hospital General Universitario Gregorio Marañón, Madrid; José Muñoz Langa, M.D., Study Chair — Hospital Universitario y Politécnico La Fe, Valencia; Alberto Carmona Bayonas, M.D., Study Chair — Hospital Universitario Morales Meseguer, Murcia; Paula Jiménez Fonseca, M.D., Study Chair — Hospital Universitario Central de Asturias, Oviedo; Pedro Pérez Segura, M.D., Study Chair — Hospital Universitario Clínico San Carlos, Madrid; Eva Martínez de Castro, M.D., Study Chair — Hospital Universitario Marqués de Valdecilla, Santander
Locations (48):
- Spain (48):
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital Universitario de Torrevieja, Elche, Alicante
  - Hospital Son Espases, Palma, Balearic Islands
  - Institut Català D'Oncologia (ICO) L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital De Sant Joan Despi Moissès Broggi, Sant Joan Despí, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital de Especialidades de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Complejo Hospitalario Univ. de Santiago, Santiago de Compostela, La Coruña
  - Hospital de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Infanta Cristina, Parla, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Complejo Hospitalario Universitario de A Coruña, A Coruña
  - Hospital Universitario San Juan de Alicante, Alicante
  - Hospital Univesitario Torrecárdenas, Almería
  - Complejo Hospitalario Universitario de Badajoz, Badajoz
  - Hospital Clínic Barcelona, Barcelona
  - Hospital de Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario San Pedro de Alcántara, Cáceres
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Virgen de la Luz, Cuenca
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitari Dr. Josep Trueta/Institut Català D'Oncología Girona, Girona
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Central de la Defensa Gómez Ulla, Madrid
  - Hospital Fundación Jimenez Díaz, Madrid
  - Hospital MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario la Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes
  - Oncoavanze, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Álvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: Undecided